CLINICAL TRIAL: NCT06041464
Title: Isolation of Cultures of Epithelial Tumor Cells and Cancer-associated Fibroblasts (CAF) From Primary Squamous Cell Carcinoma of the Head and Neck and Study of HLA-DR Expression
Brief Title: Study of HLA-DR in Cell Cultures Isolated From Primary Squamous Cell Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 3740
Record Dates: First submitted 2023-02-07; First posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2022-09

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck; Cancer
Keywords: HEAD AND NECK; CANCER; IMMUNOLOGY
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Neoplasms | interventions — Cell Culture Techniques

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Epithelial cells from healthy biopsy and tumor epithelial cells from tumor biopsy maintained in culture with: DMEM High Glucose + HAM'S F12 1:1, FBS 10%, penicillin-streptomycin 1%, L-glutamine 1%, insulin 10µg /ml, EGF 20ng/ml, Hydrocortisone 0.5µg/ml;
  • Fibroblasts from healthy biopsy and tumor associated fibroblasts (CAF) from tumor biopsy maintained in culture with: DMEM High Glucose, FBS 10%, penicillin-streptomycin 1%, L-glutamine 1%. Both fibroblasts and CAFs will be isolated from epithelial and tumor cell cultures, respectively, with a series of passages in trypsin-EDTA 0.25%
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cancer epithelial cell: cancer epithelial cells culture
  Interventions: Other: cell culture
- cancer fibroblast culture: cancer fibroblast cells culture
  Interventions: Other: cell culture

INTERVENTIONS:
Other: cell culture — isolation of cell culture
  Other Names: immunohistochemical detection

SUMMARY:
In our previous study (title: Expression of Major Histocompatibility Complex Molecules class II- HLA-DR in Squamous Cell Carcinoma of the Head and Neck. ID 2222)the Authors verified that the epithelial cells of squamous cell carcinoma of the head and neck acquire the ability to express HLA-DR. Although the role of the expression of these molecules on neoplastic cells still remains controversial, a positive association between HLA-DR expression and clinical outcome was observed by us in analogy to what was reported by several studies on various types of tumors : in squamous cell carcinoma of the larynx, colorectal cancer , stomach cancer and others. In these tumors the expression of HLA-DR correlates with the presence of immune cells such as CD16+/CD11c macrophage myeloid cells, associated with a good prognosis and T cells which, recalled in the damaged tissue, they determine the formation of an immunogenic microenvironment that could support an anti-tumor immune response. Oncology studies are in fact focusing on the role of the tumor microenvironment which is characterized by different cell populations, among which the most abundant population is represented by tumor-associated fibroblasts (CAF). CAFs are fibroblasts which, in a tumor context, assume a phenotype similar to that of myo-fibroblasts and are distinguishable from normal fibroblasts by a greater expression of α-sma, FAP and FSP-1, which represent their specific markers, as well as a greater expression of vimentin, fibronectin, and type XI collagen. Numerous evidences in different types of tumors have reported both the immunosuppressive role, as these cells are capable in vitro of inhibiting the proliferation of T lymphocytes, to favor their apoptosis or to induce the phenotype of regulatory T lymphocytes; and the pro-tumor role, as they are capable of promoting tumor proliferation and invasion, angiogenesis and metastasis, thus contributing to the worsening of the prognosis. Many studies are directing their research on which factors secreted by CAFs are responsible for their function. In particular, among the many factors secreted by CAFs, there are the interleukins IL-17 and IL-33 which, as it has been demonstrated, can induce the activation of HLA-DR molecules on bone marrow-derived mesenchymal cells . It therefore seems interesting to investigate the role of HLA-DR in relation to the presence of the tumor microenvironment represented by CAFs.

DETAILED DESCRIPTION:
Several studies have demonstrated a correlation between the expression on tumor cells of MHC II (major histocompatibility complex class II) molecules, in particular of HLA-DR (human luekocyte antigen) molecules, and the clinical outcome of the disease. Indeed, it has been observed that tumor cells under inflammatory stimulation of IFN-γ become capable of expressing MHC II molecules functioning as non-professional APCs (antigen presenting cells). The APC cells are responsible for presenting the antigen to the T lymphocytes, thus inducing their activation, which necessarily requires the presence of two signals: the first induced by the MHC molecules (MHC class II for CD4+ lymphocytes) and the second induced by Costimulatory molecules CD80 or CD86, without which lymphocytes undergo a state of anergy.

Although the role of the expression of these molecules on neoplastic cells still remains highly controversial, a positive association between HLA-DR expression and clinical outcome has been reported by several studies on various types of tumors: in squamous cell carcinoma of the larynx , colorectal cancer , stomach cancer , and others. Also in our study "Expression of the Molecules of the Major Histocompatibility Complex class II-HLA-DR in Squamous Cell Carcinoma of the Head and Neck" (ID 2222) the investigators were able to verify that the neoplastic epithelial cells of squamous cell carcinoma of the head and neck acquire the ability to express HLA-DR (data not shown, in progress of the scientific work to be presented to journal with impact factor and of the final PhD thesis in Neuroscience of the PhD student Chiara Prampolini). In some types of tumors, the expression of HLA-DR correlates with the presence of immune cells such as CD16+/CD11c macrophage myeloid cells, associated with a good prognosis and T cells which, recalled in damaged tissue, thus determine the formation of an immunogenic microenvironment which could thus support an anti-tumor immune response . Therefore, the variability in the expression of HLA-DR molecules would explain the different immune involvement in the tumor site and would condition the host's ability to stem tumor progression.

A fundamental role in tumor progression is the microenvironment, on which more and more studies are focusing. The tumor microenvironment is characterized by different cell populations, among which the most abundant population is represented by tumor-associated fibroblasts (CAF). CAFs are fibroblasts which, in a tumor context, assume a phenotype similar to that of myo-fibroblasts and are distinguishable from normal fibroblasts by a greater expression of α-sma, FAP and FSP-1, which represent their specific markers, as well as a greater expression of vimentin, fibronectin, and type XI collagen. Numerous evidences in different types of tumors have reported both the immunosuppressive role, as these cells are capable in vitro of inhibiting the proliferation of T lymphocytes, to favor their apoptosis or to induce the phenotype of regulatory T lymphocytes; and the pro-tumor role, as they are capable of promoting tumor proliferation and invasion, angiogenesis and metastasis, thus contributing to the worsening of the prognosis.

Many studies are directing their research on which factors secreted by CAFs are responsible for their function. In particular, among the many factors secreted by CAFs, there are the interleukins IL-17 and IL-33 which, as it has been demonstrated, can induce the activation of HLA-DR molecules on bone marrow-derived mesenchymal cells . It therefore seems interesting to investigate the role of HLA-DR in relation to the presence of the tumor microenvironment represented by CAFs. of the study OBJECTIVES OF THE STUDY Primary objective of the study

* Isolate tumor epithelial and cancer-associated fibroblast (CAF) cell cultures from pathological and healthy tissue samples from patients with primary squamous cell carcinoma of the head and neck Secondary objectives of the study
* To investigate the expression of HLA-DR in the obtained cell cultures. Enrolled patients and enrollment methods Calculation of the sample size The calculation of the sample size was carried out using Power Analysis, deeming acceptable a first type error equal to 5% with a test power of 90%, therefore a second type error of 10%. To determine the delta, the minimum acceptable difference to be detected between the two groups being compared (group A: healthy tissue; group B: pathological tissue) and the standard deviation relating to the populations under examination, the calculations of the effect size were followed guidelines proposed by Choen .

Patients Four patients with primary squamous cell carcinoma of the head and neck admitted for surgical treatment at the Otolaryngology Clinic, Fondazione Policlinico Gemelli, IRCCS, Rome, in the year 2020-2021 will be included in the study.

Of the 4 cases considered will be available:

* Clinical data
* Informed consent
* Tumor tissue sample
* Non-tumor tissue sample taken from material surgically removed during surgery

Informed consent The subjects involved in the study will be invited to read the project information sheet and to personally sign the informed consent for the use of their stored biological material and clinical data for research purposes.

Organic material For each patient included in the study, a biopsy will be taken both from the pathological tissue and from the healthy tissue removed during the therapeutic surgery, used as a control. Both biopsies will be cultured.

5. Study design The study is a non-profit, single-centre that consists of two phases. The expected duration of the study is 12 months.

I PHASE:

Selection of cell populations

Through specific culture media will be selected:

* Epithelial cells from healthy biopsy and tumor epithelial cells from tumor biopsy maintained in culture with: DMEM High Glucose + HAM'S F12 1:1, FBS 10%, penicillin-streptomycin 1%, L-glutamine 1%, insulin 10µg /ml, EGF 20ng/ml, Hydrocortisone 0.5µg/ml;
* Fibroblasts from healthy biopsy and tumor associated fibroblasts (CAF) from tumor biopsy maintained in culture with: DMEM High Glucose, FBS 10%, penicillin-streptomycin 1%, L-glutamine 1%. Both fibroblasts and CAFs will be isolated from epithelial and tumor cell cultures, respectively, with a series of passages in trypsin-EDTA 0.25%

Cell populations from the healthy biopsy (healthy epithelial cells and fibroblasts) will be used as negative control.

PHASE II: Evaluation of HLA-DR expression in tumor epithelial cells and tumor CAFs HLA-DR positivity will be evaluated by double immunofluorescence analysis with the addition of an epithelial marker (cytokeratin), in addition to the evaluation of the presence of classical costimulatory molecules (CD80, CD86).

HLA-DR+ tumor cells that do not express the costimulatory molecules will be stimulated in culture with the administration of IFN-ɣ and LPS, in order to induce their expression .

Statistic analysis Comparisons between categorical data (healthy and pathological tissue) will be made by chi-square test or Fisher's exact test, where appropriate. All tests will be two-tailed and an alpha <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of primary squamous cell carcinoma of the head and neck, 2) signing of informed consent for study involvement.

Exclusion Criteria:

1) patients diagnosed with non-primary squamous cell carcinoma of the head and neck and already undergoing radiotherapy, chemotherapy and immunotherapy, biological therapy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The calculation of the sample size was carried out using Power Analysis, deeming acceptable a first type error equal to 5% with a test power of 90%, therefore a second type error of 10%.
  patients Four patients with primary squamous cell carcinoma of the head and neck admitted for surgical treatment at the Otolaryngology Clinic, Fondazione Policlinico Gemelli, IRCCS, Rome, in the year 2020-2021 will be included in the study.
  Of the 4 cases considered will be available:
  * Clinical data
  * Informed consent
  * Tumor tissue sample
  * Non-tumor tissue sample taken from material surgically removed during surgery
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2023-10-02 (Estimated); Study Completion 2024-03-02 (Estimated)

PRIMARY OUTCOMES:
NUMBER OF FLASKS OF HUMAN HEALTHY TISSUE CELL CULTURE FROM THE HEALTHY HEALTHY BIOPSY BIOPSY | FROM THE DATA OF HEALTHY EPITHELIAL CELLS AND FIBROBLASTS BIOPSY UNTIL THE DATE OF CELL COLTURE ISOLATION ASSESSED UP TO 4 WEEKS
NUMBER OF FLASKS OF TUMOR ASSOCIATED EPITHELIAL CELL AND FIBROBLASTS ASSOCIATED CANCER CULTURE FROM TUMOR BIOPSY | FROM THE DATA OF TUMOR EPITHELIAL CELLS AND FIBROBLASTS BIOPSY UNTIL THE DATE OF CELL COLTURE ISOLATION ASSESSED UP TO 4 WEEKS

SECONDARY OUTCOMES:
ZERO UP TO 4 SCALE (NEGATIVE UP TO VERY INTENSIVE) IMMUNOHISTOCHEMICAL HLA-DR POSITIVITY IN HEALTHY EPITELIAL CELLS AND FIBROBLASTS CULTURES | FROM LAST ENROLLED PATIENT CELL COLTURES ISOLATION UP TO 16 WEEKS
ZERO UP TO 4 SCALE (NEGATIVE UP TO VERY INTENSIVE) IMMUNOHISTOCHEMICAL HLA-DR POSITIVITY IN TUMOR EPITELIAL CELLS AND FIBROBLASTS CULTURES | FROM LAST ENROLLED PATIENT CELL COLTURES ISOLATION UP TO 16 WEEKS

CONTACTS AND LOCATIONS:
Overall Officials: gabriella cadoni, Prof, Principal Investigator — FONDAZIONE POLICLINICO UNIVERSITARIO GEMELLI, IRCCS
Locations (1):
- Fondazione Policlinico Universitario Gemelli, Irccs, Rome, Lazio, Italy

IPD SHARING:
Plan to Share IPD: No